CLINICAL TRIAL: NCT06896903
Title: Analysis of Coronary Reactivity Testing With and Without Intracoronary Nitrate Testing
Acronym: CRT-NITRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 025-193
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-03

CONDITIONS: ANOCA - Angina With Non-obstructive Coronary Arteries; INOCA (Ischemia With Non Obstructive Coronary Artery Disease)
Keywords: Coronary Reactivity Testing; Intracoronary Nitroglycerine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Coronary Reactivity Testing with and without intracoronary nitroglycerine (Experimental): CRT will be performed in the left anterior descending and right coronary arteries. The following measures will be obtained in each of the coronaries first without intracoronary nitrates followed by a dose of 200-500 mcg of intracoronary nitrates and repeat measurements:
  * Coronary flow reserve (CFR) (normal > 2.0)
  * Index of microvascular resistance (IMR) (normal <25)
  * Resting ratio of distal coronary pressure to aortic pressure (Pd/Pa) (normal < 0.91)
  * Resting and hyperemic (using intravenous adenosine) transit time (Tm)
  * Resting full-cycle ratio (RFR)
  * Hyperemic (using intravenous adenosine) fractional flow reserve (FFR)
  * Resistive reserve ratio (RRR)
  Interventions: Diagnostic Test: Coronary reactivity testing with and without nitrates

INTERVENTIONS:
Diagnostic Test: Coronary reactivity testing with and without nitrates — CRT will be performed in the left and right coronary arteries. Measurements will be obtained in each of the coronaries first without intracoronary nitrates followed by a dose of 200-500 mcg of intracoronary nitrates and repeat measurements.

SUMMARY:
This single-arm, multi-center, prospective study will assess the coronary flow reserve (CFR), index of microcirculatory resistance (IMR), and determinants thereof (transit time, Pa, Pd) in patients before and after intracoronary nitroglycerine.

DETAILED DESCRIPTION:
This will be a single arm, multi-center, prospective interventional study. We will approach, consent, and enroll patients referred to the cardiac catheterization laboratory for coronary angiography for the indication of angina without obstructive coronary artery disease (CAD; lesions <50%, fractional flow reserve (FFR) >0.80, or non-hyperemic pressure index (RFR) <0.89). Patients will undergo invasive assessment with CRT first without IC nitrates followed by a dose of 200-500 mcg of intracoronary nitrates and repeat CRT.

Approximately 50 patients undergoing coronary angiography for evaluation of ANOCA or INOCA will be consented for this study.

The primary outcome will be comparing the variables assessed by CRT with the primary outcome being CFR before and after nitroglycerin administration.

The secondary outcomes will be IMR, Pd, Pa, RRR, and transit times before and after nitrates.

These variables will be compared to one another using paired t-tests and generalized estimating equations.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or older
2. Patient being evaluated for ANOCA or INOCA
3. Clinical suspicion for angina
4. Patient should be able to comply with the protocol.
5. Provide written informed consent before study participation.

Exclusion Criteria:

1. Existing coronary artery disease
2. Previous percutaneous interventions within the coronaries
3. Current use (within 48 hours) of long-acting nitrate therapies
4. Current use (within 48 hours) of PDE-5 inhibitors (sildenafil, tadalafil)
5. Any other condition or co-morbidity which, in the opinion of the investigator or operator, may pose a significant hazard to the subject if he or she is enrolled in the study.
6. Children below 18 years, prisoners, pregnant people and patients who are unable to provide consent are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of CFR by CRT before and after nitrates | Intra op
  The primary outcome will be comparing the variables assessed by CRT with the primary outcome being CFR before and after nitroglycerin administration.

SECONDARY OUTCOMES:
IMR, HMR, Pd/Pa, RRR, RFR, and transit times before and after nitrates. | Intra op
  The secondary outcomes will be IMR, Pd, Pa, RRR, and transit times before and after nitrates.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White The Heart Hospital - Plano, Plano, Texas, United States

REFERENCES:
- [Background] Smilowitz NR, Prasad M, Widmer RJ, Toleva O, Quesada O, Sutton NR, Lerman A, Reynolds HR, Kesarwani M, Savage MP, Sweeny JM, Janaszek KB, Barseghian El-Farra A, Holoshitz N, Park K, Albadri A, Blair JA, Jeremias A, Kearney KE, Kobayashi Y, Miner SES, Samuels BA, Shah SM, Taqueti VR, Wei J, Fearon WF, Moses JW, Henry TD, Tremmel JA; Microvascular Network (MVN). Comprehensive Management of ANOCA, Part 2-Program Development, Treatment, and Research Initiatives: JACC State-of-the-Art Review. J Am Coll Cardiol. 2023 Sep 19;82(12):1264-1279. doi: 10.1016/j.jacc.2023.06.044. PMID 37704316
- [Background] Samuels BA, Shah SM, Widmer RJ, Kobayashi Y, Miner SES, Taqueti VR, Jeremias A, Albadri A, Blair JA, Kearney KE, Wei J, Park K, Barseghian El-Farra A, Holoshitz N, Janaszek KB, Kesarwani M, Lerman A, Prasad M, Quesada O, Reynolds HR, Savage MP, Smilowitz NR, Sutton NR, Sweeny JM, Toleva O, Henry TD, Moses JW, Fearon WF, Tremmel JA; Microvascular Network (MVN). Comprehensive Management of ANOCA, Part 1-Definition, Patient Population, and Diagnosis: JACC State-of-the-Art Review. J Am Coll Cardiol. 2023 Sep 19;82(12):1245-1263. doi: 10.1016/j.jacc.2023.06.043. PMID 37704315
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439